CLINICAL TRIAL: NCT04501536
Title: Determining Optimal Treatment Intensity for Children With Language Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Mary Beth Schmitt, Assistant Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-09-0029
Record Dates: First submitted 2020-07-29; First posted 2020-08-06 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Language Impairment
Keywords: Dose; Frequency; Vocabulary; Treatment Intensity; Intensity
MeSH Terms: conditions — Language Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Frequency (Experimental): Participants will receive therapy 4 times a week for 10 weeks for 30 minutes per session.
  Interventions: Behavioral: Word Learning Intervention
- Low Frequency (Experimental): Participants will receive therapy 1 time a week for 10 weeks for 2 hours per session.
  Interventions: Behavioral: Word Learning Intervention

INTERVENTIONS:
Behavioral: Word Learning Intervention — The word learning intervention uses the 10 commercially available children's books and 6 target vocabulary words from each book that meet common criteria for appropriate vocabulary targets. Children will receive 1-on-1 treatment sessions with a trained, speech-language research assistant. Each week, 2 of 10 storybooks chosen for the study will be read with 3 of 6 targeted vocabulary words targeted from each book. The book and words targeted will be consistent between random assignment conditions. For each book reading, speech-language interns will implement word learning strategies during pre reading, during reading, and post reading. Strategies include providing a definition, a synonym, and a contextual sentence. The number of strategies used will vary on which word is being targeted; all words will be randomly assigned to a particular dose, ranging from 0 (no strategies) to 20 (all of the strategies at each reading).

SUMMARY:
The purpose of this study is to determine the amount of speech-language intervention children with language impairment need to make vocabulary gains. The investigators hope to identify the optimal amount of intervention needed as well as the point at which adding more intervention is no longer beneficial.

Participants will be randomly assigned (like a flip of a coin) to attend therapy either one time a week for 10 weeks (2 hours a session) or 4 times a week for 10 weeks (30 min per session). Each therapy session will follow a word learning intervention that is designed to increase children's word learning abilities using rich, robust word learning strategies within story book readings.

The optimal amount of intervention relates to duration, dose, and frequency. Duration refers to how long the child is seen for (e.g., 10 weeks, 1 year). Dose represents the number of exposures to each new vocabulary word within a therapy session. Frequency represents the number of therapy sessions per week.

The investigators will test the hypothesis that distributed learning leads to higher gains. The investigators propose that the greatest gains will be observed for children who receive high-frequency/low-dose or low-frequency/high-dose treatments as compared to children who receive high-frequency/high-dose or low-frequency/low-dose treatments.

The investigators will test the hypothesis that for both low-frequency and high-frequency treatments, there is a point at which increases in treatment dose do not correspond to any additional gains in children's vocabulary skills during treatment.

At the close of this four-year study, evidence concerning optimal treatment intensity of a word learning intervention will be instrumental for immediately informing speech-language pathologists in how much vocabulary treatment to prescribe as well as for designing additional clinical trials by our and other research teams.

DETAILED DESCRIPTION:
The purpose of this study is to determine the optimal treatment intensity of a word learning intervention for improved measures of vocabulary immediately post intervention and at 6-months follow up by addressing 3 specific aims.

1. to determine whether low frequency (massed) or high frequency (distributed) conditions are more effective intervention schedules with respect to children's vocabulary gains during treatment. Using a causally interpretable research design with children randomly assigned to both conditions, the investigators will test the hypothesis that high frequency treatment will be more effective than low frequency schedules, informed from our own research as well as that proposed by distributed learning theorists. The investigators propose that the greatest gains will be observed immediately post intervention as well as 6-months post intervention for children who receive high-frequency treatment as compared to children who receive low-frequency treatment.
2. to determine the optimal number of dose exposures within each condition of frequency. Using a causally interpretable research design, with planned variations in dose, the investigators will test the hypothesis that increases in dose are beneficial when treatment frequency is low, and similarly that low levels of dose are beneficial when frequency is high. The investigators propose that the greatest gains will be observed for children who receive high-frequency/low-dose or low-frequency/high-dose treatments as compared to children who receive high-frequency/high-dose or low-frequency/low-dose treatments.
3. to identify thresholds of cumulative intensity after which additional exposures provide no additional benefit to children's vocabulary gains, corresponding to a point of 'diminishing returns'. The investigators will test the hypothesis that for both low-frequency and high-frequency treatments, there is a point at which increases in treatment dose do not correspond to any additional gains in children's vocabulary skills during treatment.

The proposed study features a two-group pre/post experimental design with random assignment to target words across six dose exposures. Using blocked random assignment, each child will first be randomized to a low-or high-frequency treatment condition. Target words will then be randomly assigned to one of six dose exposures (0, 4, 8, 12, 16, 20 with 0 serving as a control). Thus, this study will measure both between child (frequency) and within child (dose) variance attributed to intensity of treatment. Children who meet all eligibility criteria and are enrolled in the study will be randomly assigned to one of the two conditions, high-or low-frequency, as previously described.

Each child will receive one-on-one treatment sessions each week for 10 weeks according to their assigned frequency (one or four sessions per week for a total of 10 or 40 sessions, respectively) over the summer period. Each session will follow an efficacious word learning intervention. The word learning intervention uses the 10 commercially available children's books from previous studies. Each week, 2 of the 10 storybooks will be read, with 3 of the 6 vocabulary words targeted from each book. The book and words targeted will be consistent between frequency conditions. For the high-frequency condition, each book will be read once per session across 4 sessions, for a total of 4 readings per book each week. For the low-frequency condition, each book will be read 4 times in 1 session for a total of 4 readings per book each week, thereby keeping the number of book-readings equal across conditions. Over the course of the 10-week intervention, two books will be read each week and all 10 books will be read twice throughout the intervention. Three of the 6 targeted words will be taught the first week the book is read and the other 3 of 6 targeted words taught the second week the book is read. Each child will receive a total of 120 minutes of therapy each week, which equates to 14-16 hours of therapy (approximately 4 hours of therapy per day for 4 days).

The word learning intervention is designed to increase children's word learning abilities using rich, robust word learning strategies within story book readings including provision of a synonym (e.g., A furnace is like a heater), definition (e.g., Furnace means something used to make heat to warm buildings), and context sentence (e.g., Today it was cold outside so mom turned on the furnace) during pre-book reading, book reading, and post-book reading activities. During the pre-book reading, the intern will discuss the target words that the child will hear in the book, with the exception of the word assigned to the 0 exposure condition. During this portion of the intervention, the speech-language intern will use zero, one or two strategies, depending on the assigned dose. During the book reading portion of the intervention, the intern will read the book in its entirety. The intern will either not elaborate the target word (0 dose) or will offer a synonym as the word is read in the book. During the post-book reading, the intern will use zero, one, or two strategies depending on the assigned dose.

ELIGIBILITY:
Inclusion Criteria:

* Is between the ages of 5:0-8:11
* Has a primary diagnosis of a language impairment with deficits in vocabulary
* Primarily communicates in English
* Scores at or below 10th percentile on at least one of these three vocabulary assessments:

  1. Semantics subtest of the Diagnostic Evaluation of Language Variation (DELV)
  2. Vocabulary subtests of the Test of Language Development (TOLD-P:5); or
  3. Comprehensive Receptive and Expressive Vocabulary (CREVT)

Exclusion Criteria:

* Children with concomitant diagnoses that may underlie observed language difficulties (e.g., autism, hearing loss, severe cognitive disability)

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Definition Task | Within 2 weeks of the last intervention session
  The definition task assesses children's abilities to define the 60 intervention target words. To administer the definition task, children are shown a picture representing each targeted word and asked to define it.
Generalized Change in Definition Task | 6 months after the last intervention session
  The definition task assesses children's abilities to define the 60 intervention target words. To administer the definition task, children are shown a picture representing each targeted word and asked to define it.

SECONDARY OUTCOMES:
Change in Word Definition Task Expressive One-Word Picture Vocabulary Test -Fourth Edition (EOWPVT-4); Standardized | Within 2 weeks of the last intervention session
  The EOWPVT-4 is an individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures.
Generalized Change in Word Definition Task Expressive One-Word Picture Vocabulary Test -Fourth Edition (EOWPVT-4); Standardized | 6 months after the last intervention session
  The EOWPVT-4 is an individually administered, norm-referenced assessment of how well a person can name objects, actions, or concepts presented in full-color pictures.
Change in Receptive One-Word Picture Vocabulary Test-Fourth Edition (ROWPVT-4); Standardized | Within 2 weeks of the last intervention session
  The ROWPVT-4 is an individually administered, norm-referenced assessment of how well a person can match a word that is heard to objects, actions, or concepts presented in pictures.
Generalized Change in Receptive One-Word Picture Vocabulary Test-Fourth Edition (ROWPVT-4); Standardized | 6 months after the last intervention session
  The ROWPVT-4 is an individually administered, norm-referenced assessment of how well a person can match a word that is heard to objects, actions, or concepts presented in pictures.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Beth Schmitt, PhD, Principal Investigator — The University of Texas at Austin; Laura Justice, PhD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - University of Texas at Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
We would not release protected information specific to individual participants, but will share de-identified study data and protocols with other researchers who could use the data to advance knowledge of treatment processes for children with language impairment.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data and supporting information will be available one year after the study completion (1/31/2025) for 5 years.
Access Criteria: Researchers interested in our data or supporting documents should contact the PI: Dr. Mary Beth Schmitt (see contact information)

DOCUMENTS (1):
  • Informed Consent Form (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT04501536/ICF_001.pdf